CLINICAL TRIAL: NCT01494753
Title: Pharmacokinetics, Efficacy and Safety Assessment of T2345 Compared With Active Comparator in Newly Diagnosed Patients With Open-angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: LT2345-PII-10/07(IN)
Record Dates: First submitted 2011-12-08; First posted 2011-12-19 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Primary Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Prostaglandins

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Prostaglandin (Active Comparator): One drop.
  Interventions: Drug: Prostaglandin
- T2345 (Experimental): One drop
  Interventions: Drug: T2345

INTERVENTIONS:
Drug: T2345 — One drop at 8.00pm.
  Arms: T2345
Drug: Prostaglandin — One drop at 8.00pm.
  Arms: Prostaglandin

SUMMARY:
The purpose of this study is to assess the pharmacokinetics, efficacy and safety of T2345 versus an active comparator.

ELIGIBILITY:
Inclusion Criteria:

* Untreated bilateral newly diagnosed patients with primary open angle glaucoma

Exclusion Criteria:

* Any ocular hypertension other than chronic open angle glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

REFERENCES:
- [Derived] Aptel F, Choudhry R, Stalmans I. Preservative-free versus preserved latanoprost eye drops in patients with open-angle glaucoma or ocular hypertension. Curr Med Res Opin. 2016 Aug;32(8):1457-63. doi: 10.1080/03007995.2016.1202818. Epub 2016 Jun 25. PMID 27310103

RESULTS

PARTICIPANT FLOW:
Groups:
- Prostaglandin/T2345; T2345/Prostaglandin: One drop at 8.00pm.
Period: Day0-Day42
Arm/Group | Prostaglandin/T2345 | T2345/Prostaglandin
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Day42-Day84
Arm/Group | Prostaglandin/T2345 | T2345/Prostaglandin
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prostaglandin/T2345 | T2345/Prostaglandin | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (12.6) | 50.2 (13.4) | 50.7 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 13 | 8 | 21
Region of Enrollment [Number; unit: participants]
  India | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Mean Intra Ocular Pressure (IOP) at 8.00am
Description: Efficacy criteria at 8.00am on Day 42 and on Day84. Worse Eye= the eligible eye (with at least one out of the 4 individual IOP values on Day 0 >= 22 and <=30mmHg) with the highest individual IOP at 8.00am on Day 0. If both eyes are eligible and have the same individual IOP at 8.00am on Day 0, the right eye is considered.
Time Frame: Day 42 and Day 84 (8.00am for the IOP)
Population: Per protocol (PP) set: All patients enrolled in the study for whom any follow-up efficacy information was evaluable and who did not show any major protocol deviation that could affect the efficacy assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Prostaglandin/T2345 | T2345/Prostaglandin
Number analyzed (Participants) | 15 | 15
mmHg
  IOP at 8am for the worse eye (PPset) D42 | 16.6 (3) | 16.3 (2.3)
  IOP at 8am for the worse eye (PPset) D84 | 17 (2.2) | 15.7 (2.9)

ADVERSE EVENTS:
Arm/Group | Prostaglandin | T2345
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prostaglandin (N=30) | T2345 (N=30)
Status Asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the results of the Trial are the sole and exclusive property of THEA, and cannot be used in whatever form without prior written agreement of THEA.